CLINICAL TRIAL: NCT07219771
Title: A Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm, Phase 3 Study of Intra-Articular Administration of an Allogeneic Human Placental Tissue Particulate (PTP-001) for the Treatment of Knee Osteoarthritis
Brief Title: A Study to Evaluate the Efficacy and Safey of PTP-001 (MOTYS™) in Knee Osteoarthritis Patients
Acronym: MOTION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Doron Therapeutics Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOA-25-03
Record Dates: First submitted 2025-10-21; First posted 2025-10-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded trial, in which neither participant nor investigator will know the content of the investigational product. Additionally, unblinded personnel that prepare the syringe and administer the injection must not be involved in any other operational aspects of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTP-001 200 mg (Experimental): A single intra-articular injection in the target knee of PTP-001 200 mg
  Interventions: Biological: PTP-01
- Placebo / saline vehicle (Placebo Comparator): A single intra-articular injection in the target knee of 4 mL of placebo control (0.9% sodium chloride injection, USP)
  Interventions: Other: Placebo control / saline vehicle

INTERVENTIONS:
Biological: PTP-01 — Allogeneic human placental tissue particulate (PTP-001) is administered as a single intra-articular injection to the target knee after resuspension with saline.
  Other Names: MOTYS™; allogeneic human placental tissue particulate
  Arms: PTP-001 200 mg
Other: Placebo control / saline vehicle — The placebo control, physiological saline (0.9% sodium chloride injection, USP), is administered as an intra-articular injection to the target knee.
  Other Names: Normal saline; Physiological saline
  Arms: Placebo / saline vehicle

SUMMARY:
This is a multicenter, prospective, randomized, double-blind, placebo-controlled, parallel-arm, Phase 3 study of intra-articular administration of PTP-001 (MOTYS) for the treatment of knee osteoarthritis.

The purpose of the trial is to evaluate the efficacy, safety, and tolerability of a single intra-articular injection of PTP-001 compared to placebo over a 52-week period in participants with radiographic and symptomatic knee OA.

DETAILED DESCRIPTION:
The participants will be randomized in a 1:1 ratio to receive one of either PTP-001 or placebo injection. Each participant will be administered a single dose of investigational product (IP) (active or placebo) on Day 1.

The trial will consist of a Screening period (up to 28 days prior to treatment), a treatment phase (1 day) and a follow-up phase (12 months following treatment). A total of at least 260 participants are planned to be randomized (130 participants/group).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 40 to 80 years.
2. Presenting with symptomatic knee OA with Kellgren-Lawrence (KL) radiographic classification of 2 or 3 (mild or moderate), as assessed by the central reading facility.
3. Primary source of pain throughout the body is due to OA in the target knee.
4. Target knee pain ≥ 20 and ≤ 40 out of 50 on the WOMAC® numerical rating scale (NRS) 3.1 pain questionnaire (sum of 5 questions) at Screening and Baseline.
5. Onset of symptomatic OA of the target knee was at least 6 months prior to Screening.
6. Insufficient, failed response, or intolerance to analgesics and / or non-steroidal anti-inflammatory drugs (NSAIDs), as reported by the participant.
7. If female, must meet all of the following:

   1. Not breast feeding,
   2. Not planning to become pregnant during the study,
   3. Must abstain from ova / egg donation during the study,
   4. If of childbearing potential, must have a negative pregnancy test result within 72 hours prior to receiving the intra-articular injection, and must commit to the use of a highly effective form of birth control for at least 90 days after the injection.
8. Willing to remain on the same oral "rescue" (as needed) analgesic as the only pharmacologic treatment for knee pain during the study.
9. Willing to abstain from taking any illicit or unauthorized medications for treatment of OA or any other concurrent condition during the study.
10. Willing to comply with post-injection restrictions.
11. Written informed consent is obtained from the participant.

Exclusion Criteria:

1. Participant is non-ambulatory (unable to walk > 50 feet / 15 meters without assistance).
2. Clinically severe obesity as defined by the National Institutes of Health (body mass index ≥ 40 kg/m2) at Screening and / or Baseline.
3. Contralateral (non-target) knee pain is ≥ 6 out of 50 on the WOMAC® NRS 3.1 pain questionnaire (sum of 5 questions) at Screening or at Baseline.
4. At Baseline, difference between the first and second WOMAC pain scores is ≥ 3 for the target knee.
5. Contralateral (non-target) knee pain is experienced for ≥ 14 days in the month.
6. Use of any analgesia during the washout period (5 half-lives) at Screening or Baseline.
7. Participation in any investigational study within 30 days (or 5 half-lives, whichever is longer) prior to Screening or planning to participate in any other investigational drug or device clinical trials within 30 days of study completion.
8. Currently requires use of a lower extremity prosthesis and / or a structural knee brace (ie, a knee brace that contains hardware).
9. Clinically significant effusion of the target knee at either the Screening or Baseline visits as determined by physical examination (eg, ballotable patella or positive bulge sign).

   Note: Participants presenting with effusion may be enrolled in the study after undergoing knee aspiration to remove excess fluid in the target joint.
10. Severe (excessive) malalignment of the tibial-femoral axis assessed radiographically (by previous X-ray, rather than that performed for Kellgren-Lawrence assessment).
11. Presence of active infection in the target knee or systemic infection requiring treatment within the 3 months prior to Screening.
12. Clinical diagnosis of inflammatory arthritis (eg, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, etc.) established by clinical history, examination, or serology.
13. Participant is receiving, has received, or plans to receive any of the following therapies:

    1. Prior administration of hyaluronic acid, extended-release corticosteroid (eg, Zilretta®), platelet-rich plasma (PRP), or stem cell therapies by intra-articular injection(s) of the target knee within 6 months prior to Screening.
    2. Prior administration of corticosteroid by intra-articular injection of the target knee within 3 months prior to Screening or into any other joint within 30 days prior to Screening.
    3. Current chronic systemic use of corticosteroids in doses exceeding the equivalent of 10 mg prednisolone daily.
    4. Treatment with any investigational therapy (drug, device, or biologic) within 3 months prior to Screening or is planned for the duration of the study.
    5. Treatment with immunosuppressive medication (not including mild transient immunosuppressants such as corticosteroids) or chemotherapy within the past 5 years.
14. Chronic use of narcotics or alcohol abuse within the past 6 months prior to Screening.
15. Surgery to either knee (including arthroscopy) within 6 months prior to receiving the intra-articular injection or planned surgery of either knee within 6 months after the injection.
16. Participant previously underwent arthroplasty of the target knee.
17. Presence of joint instability or complaints of locking, intermittent limitation in range of motion, or loose body sensation, suggestive of internal derangement of the knee (either extremity).
18. Diagnosis of lower extremity gout or pseudo-gout in the past 6 months prior to Screening.
19. History of, or current manifestation of, osteonecrosis of either knee.
20. Significant acute (within the past 3 months) injury to the target knee.
21. History of receiving a solid organ or hematologic transplant.
22. History of malignancy, radiotherapy, or chemotherapy for malignancy within the past 5 years, except for basal or squamous cell carcinoma of the skin.
23. History of prior radiation therapy of the target knee.
24. History of autoimmune disease affecting the musculoskeletal system.
25. Known (documented) history of acquired immune deficiency syndrome or human immunodeficiency virus (HIV).
26. Any condition causing pain in or around the target knee (eg, radiating pain or pain in another region of the ipsilateral lower extremity) that may interfere with assessment(s) of the target knee. 27. Other chronic pain anywhere in the body that requires the chronic use of analgesic medications, such as knee OA of the contralateral (non-target) knee, fibromyalgia, tendonitis, plantar fasciitis, neuropathic pain, lower back pain, etc.

28. Known presence of any concurrent medical condition (eg, hematologic renal, hepatic, cardiac, or coagulation abnormalities) that in the Investigator's judgment would interfere with the required study assessments and study participation.

29. Participant is involved in litigation (eg, worker's compensation) for a medical condition or injury at any anatomical site.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants meeting strict responder criteria for improvement in knee function. | 6 months
  To qualify as a "strict responder for improvement in knee function", an improvement of ≥ 50% in WOMAC Function subscale score is required, with an absolute change ≥ 20 points in the score.
Proportion of participants meeting strict responder criteria for improvement in knee pain. | 6 months
  To qualify as a "strict responder for improvement in knee pain", an improvement of ≥ 50% in WOMAC Pain subscale score is required, with an absolute change ≥ 20 points in the score.

SECONDARY OUTCOMES:
Proportion of participants meeting strict responder criteria for improvement in knee function. | 9 months and 12 months
Proportion of participants meeting strict responder criteria for improvement in knee pain. | 9 months and 12 months
Change from pretreatment Baseline in participant self-reported assessment of OA by PGA-OA score. | 6 months, 9 months, and 12 months
Change from pretreatment Baseline in participant self-reported function of the treated knee as assessed by WOMAC Function subscale score. | 6 months, 9 months, and 12 months
Change from pretreatment Baseline in participant self-reported pain at the treated knee as assessed by WOMAC Pain subscale score. | 6 months, 9 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Professor David Hunter, Principal Investigator — Chair of Rheumatology at University of Sydney and Royal North Shore Hospital
Locations (9):
- Australia (9):
  - Emeritus Research Sydney, Botany, New South Wales
  - Genesis Research Services, Broadmeadow, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - University of the Sunshine Coast Clinical Trials, Birtinya, Birtinya, Queensland
  - University of the Sunshine Coast Clinical Trials, Morayfield, Morayfield, Queensland
  - University of the Sunshine Coast Clinical Trials, Noosa, Noosaville, Queensland
  - Momentum Clinical Research Taringa, Taringa, Queensland
  - Momentum Clinical Research Wellers Hill, Tarragindi, Queensland
  - Momentum Clinical Research Sunshine, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flannery CR, Buddin KE, Begum L, Nasert MA, Catalfamo B, Semler EJ, Fortier LA. Composition and Bioactivity of a Placental Tissue Particulate (PTP-001) Indicate Greater Potential than Platelet-Rich Plasma for the Treatment of Osteoarthritis. Cartilage. 2023 Dec;14(4):467-472. doi: 10.1177/19476035231159748. Epub 2023 Mar 13. PMID 36912174
- [Result] Flannery CR, Seaman SA, Buddin KE, Nasert MA, Semler EJ, Kelley KL, Long M, Favret J, Pavesio A, Loeser RF. A novel placental tissue biologic, PTP-001, inhibits inflammatory and catabolic responses in vitro and prevents pain and cartilage degeneration in a rat model of osteoarthritis. Osteoarthritis Cartilage. 2021 Aug;29(8):1203-1212. doi: 10.1016/j.joca.2021.03.022. Epub 2021 May 20. PMID 34023528
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34023528/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36912174/